CLINICAL TRIAL: NCT01812954
Title: Economic Evaluation of Systemic Treatments for Moderate-to-severe Psoriasis
Status: Completed | Type: Observational
Sponsor: Jochen Schmitt. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jochen Schmitt., Director of Center for evidence-based healthcare, Technische Universität Dresden
Organization: Technische Universität Dresden (Other)
Other Study IDs: PSO-GOE; 50310 (Other Grant/Funding Number: MSD Sharp&Dohme GmbH)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Psoriasis
Keywords: moderate-to-severe psoriasis; cost utility analysis; cost effectiveness analysis; systemic treatment
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate; Cyclosporins; fumaric acid; Acitretin; Infliximab; Etanercept; Adalimumab; Ustekinumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methotrexate
Drug: Cyclosporins
Drug: fumaric acid
Drug: Acitretin
Drug: Infliximab
Drug: etanercept
Drug: Adalimumab
Drug: Ustekinumab

SUMMARY:
This study is health economic analysis of medicinal treatment options for moderate-to-severe psoriasis vulgaris from the societal perspective. Efficacy data and other clinical outcomes will be derived from an up-to-date meta-analysis of randomized clinical trials (RCTs) for moderate-to-severe psoriasis. Direct and indirect costs will be extracted from various different sources, including summary of product characteristics (SPCs) and the German S3 guideline on psoriasis care, health care utilization data and official statistics.

The study aims to investigate the comparative cost-effectiveness of biologic and conventional systemic treatments currently (as of June 1st, 2012) approved for moderate-to-severe plaque-type psoriasis in Germany. Effectiveness will be measured by means of the pooled (Psoriasis Area and Severity Index) PASI-75 response rates as reported in RCTs Direct cost as well as indirect cost will be considered.

ELIGIBILITY:
Inclusion Criteria:

-diagnosis of moderate-to-severe psoriasis

Exclusion Criteria:

-

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with moderate-to-severe psoriasis, who require systemic treatment to adequately control the disease
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cost per quality-adjusted life year (QALY) gained through treatment with each individual agent compared to supportive care as well as compared to placebo | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Schmitt, MD, MPH, Principal Investigator — University Dresden